CLINICAL TRIAL: NCT02564653
Title: Implementing Tobacco Use Guidelines in Community Health Centers in Vietnam Public Health System:a Rural Model
Brief Title: Implementing Tobacco Use Guidelines in Community Health Centers in Vietnam Public Health System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-01422
Record Dates: First submitted 2015-09-02; First posted 2015-10-01 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technical Assistance, training,clinical reminders (Other): provider adherence to tobacco use treatment guidelines
  Interventions: Behavioral: Technical Assistance, training and clinical reminders
- TTC + help of community health workers (Other): We will assess this secondary aim by comparing smoking cessation outcomes among smokers who receive brief provider counseling alone only vs. smokers who receive provider counseling + community health worker counseling. The purpose of this assessment is to specifically analyze the impact of the community health worker counseling component of the intervention using a quasiexperimental design that leverages the larger RCT.
  Interventions: Behavioral: TTC+Referral to Community Health Worker

INTERVENTIONS:
Behavioral: Technical Assistance, training and clinical reminders — Technical Assistance, training and clinical reminders (TTC)
  Arms: Technical Assistance, training,clinical reminders
Behavioral: TTC+Referral to Community Health Worker — TTC+ referral to a VHW for additional counseling and follow-up
  Arms: TTC + help of community health workers

SUMMARY:
Vietnam has a smoking prevalence that is the second highest among South East Asian countries (SEACs). With a population of approximately 90 million, Vietnam also has the second largest total number of adult smokers (over 16 million) in SEA. According to the World Health Organization (WHO), most reductions in mortality from tobacco use in the near future will be achieved through helping current users quit. Tobacco use treatment, as defined by the U.S. Preventive Health Service Guideline (Guideline) on Treating Tobacco use and Dependence, is evidence-based and highly cost-effective. Yet, in the U.S. and globally, adoption of recommended care is suboptimal. The objective of this proposal is to fill the current research-to-practice gap by conducting a randomized controlled trial that compares the effectiveness and cost effectiveness of two practical and highly replicable strategies for implementing evidence-based guidelines for the treatment of tobacco use in public health clinics in Vietnam. The proposed implementation strategies draw on evidence-based approaches, and the WHO's recently released guidelines for implementing Article 14 of the Framework Convention on Tobacco Control (FCTC). The FCTC is an evidence-based treaty that was developed by the WHO in response to the globalization of the tobacco epidemic. Vietnam ratified the FCTC in 2004; however, they have not taken steps to implement Article 14 which specifies the need to integrate best practices for treating tobacco use and dependence into routine preventive care. The proposed implementation strategies also build on the growing literature that supports the effectiveness of integrating community health workers as members of the health care team to improve access to preventive services.

DETAILED DESCRIPTION:
The long-term goal of the project is to develop a generalizable model for implementing evidence-based tobacco use treatment within existing health systems locally and globally. The objective of this proposal is to fill the current research-to-practice gap by conducting a randomized controlled trial that compares the effectiveness and cost of two practical and highly replicable strategies for implementing evidence-based guidelines for the treatment of tobacco use in public health clinics and community based settings in Vietnam. The proposed implementation strategies draw on evidence-based approaches and the WHO's recently released guidelines for implementing Article 14 of the Framework Convention on Tobacco Control (FCTC). The FCTC is an evidence-based treaty that was developed by the WHO in response to the globalization of the tobacco epidemic Article 14specifies the need to integrate clinical best practices for treating tobacco use and dependence into routine preventive care. The proposed implementation strategies also build on the growing literature that supports the effectiveness of integrating community health workers as members of the health care team to improve access to preventive services.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligibility:
* Current patients at community health center for routine visit
* 18 years or older
* Current or regular smoker (>1 cigarette in past 7 days)
* Willingness to complete survey
* 18 years or older
* Willingness to complete survey or interview

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4733 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Adherence to tobacco use treatment guidelines and costs | Up to 12 months
  patient exit interviews

SECONDARY OUTCOMES:
Smoking abstinence | Up to 12 months
  Surveys will be conducted in person and smoking abstinence will be validated using carbon monoxide (CO) monitoring

OTHER OUTCOMES:
Barriers and facilitators for tobacco use treatment | Up to 12 months
  practice environment checklist to inventory current policies, work flow, systems (e.g. chart systems) and staff roles and responsibilities in general and specifically related to tobacco use treatment

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, MPH, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] VanDevanter N, Vu M, Nguyen A, Nguyen T, Van Minh H, Nguyen NT, Shelley DR. A qualitative assessment of factors influencing implementation and sustainability of evidence-based tobacco use treatment in Vietnam health centers. Implement Sci. 2020 Sep 9;15(1):73. doi: 10.1186/s13012-020-01035-6. PMID 32907603
- [Derived] VanDevanter N, Kumar P, Nguyen N, Nguyen L, Nguyen T, Stillman F, Weiner B, Shelley D. Application of the Consolidated Framework for Implementation Research to assess factors that may influence implementation of tobacco use treatment guidelines in the Viet Nam public health care delivery system. Implement Sci. 2017 Feb 28;12(1):27. doi: 10.1186/s13012-017-0558-z. PMID 28241770